CLINICAL TRIAL: NCT05001620
Title: Implementation of a Telehealth Palliative Care Model for Persons With Dementia
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Joan Carpenter, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00095001; U54AG063546 (NIH)
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Palliative Care; Dementia
Keywords: Dementia; Palliative Care; Telehealth; Nursing Homes
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Consultation in Post-Acute Care (Experimental): Subjects will receive usual care plus a telehealth palliative care consultation by specialty providers who will document their findings in the Electronic Health Record (EHR), and communicate their findings and recommendations to the clinical team.
  Interventions: Other: Palliative Care Consultation
- Stakeholder Engagement (No Intervention): We will engage stakeholders in a stakeholder engagement plan that include Palliative Care providers; Social Work (SW) NH champions; post-acute care unit nursing staff and providers (including medial directors); NH leadership, information technology staff; and a PLWD and their care partners in focus groups and one on one semi structured interviews via phone or videoconference.

INTERVENTIONS:
Other: Palliative Care Consultation — The PC provider conducts the structured PCC-PAC via videoconference or telephone with the PLWD and/or their care partner and the social work (SW) champion in the NH. The SW and PC provider will set up a mutually agreed upon consultation day/time with the PLWD and/or care partner, within 5 business days of NH admission and follow up visits will occur no more than 30 days later (if needed).
  Arms: Palliative Care Consultation in Post-Acute Care

SUMMARY:
Grounded in the Reach-Effectiveness-Adoption-Implementation-Maintenance (RE-AIM) Model, this study will assess the implementation outcomes of the Nurse Practitioner (NP) delivered telehealth Palliative Care Consultation in Post-Acute Care (PCC-PAC) intervention for persons living with dementia (PLWD) and their care-partners newly admitted to nursing homes (NHs) for post-acute care.

DETAILED DESCRIPTION:
This single arm embedded pragmatic pilot clinical trial will provide data to assess the implementation outcomes of the Nurse Practitioner (NP) delivered telehealth Palliative Care Consultation in Post-Acute Care (PCC-PAC) intervention among 30 persons living with dementia (PLWD) and their care-partners newly admitted to one nursing homes (NH) for post-acute care.

ELIGIBILITY:
Inclusion Criteria:

Stakeholders:

* (1) PC provider
* (2) Social Work (SW) NH champions
* (3) post-acute care unit nursing staff and providers (including medical directors)
* (4) NH leadership, information technology staff
* (5) PLWD and their care partner(s).

Person Living with Dementia (PLWD)

* documented dementia diagnosis
* admitted for post-acute care
* age ≥ 60 years
* if unable to participate in a conversation or lacking capacity to make healthcare decisions as determined by the NH staff/providers, a care partner who can act as a surrogate decision maker in the PCC-PAC.

Exclusion Criteria:

Stakeholders:

-PLWD who receives the intervention

PLWD:

* planned discharge within 48 hours of screening
* currently receiving hospice care

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Collingswood Rehabilitation and Healthcare Center, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement
Started | 2 | 14
Completed | 1 | 14
Not Completed | 1 | 0
Not completed — Didn't complete the telehealth Palliative Care Consultation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement | Total
Number analyzed (Participants) | 2 | 14 | 16
Age, Customized [Count of Participants; unit: Participants]
  >18 years of age | 2 | 14 | 16
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 0 | 1
  Female | 0 | 0 | 0
  Unknown | 1 | 14 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 14 | 15
Region of Enrollment [Number; unit: participants]
  United States | 2 | 14 | 16

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Skilled Nursing Facility (SNF)-PCC Recommendations
Description: Investigators will determine a recommendation adherence score after each participants' encounter. Each recommendation will be assigned 2 points, then will define full (2 points), partial (1 point) and no adherence (0 point) to each recommendation. Investigators will sum the points for each SNF-PCC recommendation and use this as the denominator. Investigators will sum each recommendation with full, partial, no adherence and use this as the numerator. The fraction will be converted to a percentage ranging from 0-100% reflecting the recommendation adherence score.
Time Frame: 30 days post admission
Population: no data were collected
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Hospitalizations
Description: Number of hospitalization(s)
Time Frame: 30 days post admission
Population: The one participant that completed the study did not have any hospitalizations. The Stakeholders were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Completed Stakeholder Interviews/Focus Groups
Description: We engaged participants in focus groups and semi-structured interviews to deepen understanding of barriers and facilitators to telehealth palliative care implementation.
Time Frame: 1 year
Population: no arm 1 participants were enrolled in arm 2
Measure: Count of Participants; unit: Participants
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement
Number analyzed (Participants) | 2 | 14
Participants | 1 | 14

ADVERSE EVENTS:
Time Frame: 30 days post admission
Arm/Group | Palliative Care Consultation in Post-Acute Care | Stakeholder Engagement
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/14
Other Adverse Events (participants affected / at risk) | 0/2 | 0/14

LIMITATIONS AND CAVEATS:
Despite multiple, iterative adaptations to implementation, including recruiting new sites and clinical partners, we were unable to enroll the targeted 30 patients in the trial. Two PLWD enrolled in the clinical trial, one completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT05001620/Prot_000.pdf